CLINICAL TRIAL: NCT07118735
Title: A Standardized Extract of Cultured Lentinula Edodes Mycelia (AHCC®) as Immune Modulator in Cancer Patients Treated With Immunotherapy: a Phase 2 Double-blind, Randomized, Placebo-controlled Trial
Brief Title: AHCC® as Immune Modulator in Cancer Patients Treated With Immunotherapy
Acronym: NCKUH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-BR-114-016; NationalCheng-KungU (Registry Identifier: National Cheng-Kung University Hospital Clinical Trial Center)
Record Dates: First submitted 2025-07-11; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma
Keywords: AHCC® (Active Hexose Correlated Compound); immunotherapy; liver cancer; functional food
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Dextrins

STUDY DESIGN:
Intervention Model Description: This is a prospective double-blind, randomized, placebo-controlled trial aims to investigate whether add-on of a standardized extract of cultured Lentinula edodes mycelia (AHCC®) can enhance the effect of immunotherapy in cancer patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants receive oral administration of 3g AHCC® daily (Experimental): 3 grams of AHCC taken orally once daily until disease progression or intolerance
  Interventions: Dietary Supplement: A standardized extract of cultured Lentinula edodes mycelia (AHCC®)
- Placebo (Placebo Comparator): 3 grams of dextrin (placebo) taken orally once daily until disease progression or intolerance
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: A standardized extract of cultured Lentinula edodes mycelia (AHCC®) — 3 grams of AHCC® taken orally once daily for 6 months or until disease progression or intolerance
  Arms: participants receive oral administration of 3g AHCC® daily
Dietary Supplement: Placebo — 3 grams of dextrin (placebo) taken orally once daily for 6 months or until disease progression or intolerance
  Other Names: dextrin
  Arms: Placebo

SUMMARY:
This is a prospective, double-blind, randomized, placebo-controlled trial to evaluate whether AHCC® (Active Hexose Correlated Compound) can enhance the effect of immunotherapy in liver cancer patients.

DETAILED DESCRIPTION:
Objectives:

Assess the potential of AHCC® to improve immunotherapy outcomes Evaluate progression-free survival (PFS) Evaluate overall survival (OS) Assess safety and tolerability

Method:

Participants will take 3 grams of AHCC® or placebo orally each day Treatment will continue until disease progression, treatment intolerance or other treatment options become available.

Note:

AHCC® is a novel functional food with immune-modulating potential.

ELIGIBILITY:
Inclusion Criteria:

* 1.Liver cancer patient who will receive immunotherapy
* 2.At least one measurable tumor, according to RECIST version 1.1, that has not been treated with any local procedure.
* 3.Age >=20 years old.
* 4.ECOG performance status 0 or 1.
* 5.White blood count >=2,000/microliter ; platelet count >=60,000/microliter.
* 6.Liver transaminases (ALT and AST) <=5 times upper limit of normal values (ULN); total bilirubin <= 2 times ULN; creatinine clearance or eGFR > 50 mL/min (either Cockcroft-Gault or MDRD is acceptable, whichever is higher).
* 7.Subjects with chronic hepatitis B virus infection (HBV surface antigen (HBsAg) positive) must start antiviral therapy with nucleoside analogs (e.g., entecavir or tenofovir, according to current practice guidelines) before start of study drug treatment.

Exclusion Criteria:

* 1.Major systemic diseases that the investigator considers inappropriate for participation.
* 2.Any active autoimmune disease or history of known autoimmune disease except for vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* 3.Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* 4.Prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* 5.Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* 6.Prior organ allograft or allogeneic bone marrow transplantation.
* 7.Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as assessed by RECIST v1.1 | Every 12 weeks up to 24 months
  Tumor response will be assessed by imaging (CT scan preferred) every 12 weeks using RECIST version 1.1 criteria. Objective Response Rate (ORR) is defined as the proportion of participants achieving a Complete Response (CR) or Partial Response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by RECIST v1.1 | Up to 24 months
  PFS is defined as the time from the start of treatment to the first documentation of disease progression or death from any cause, whichever occurs first. Tumor response will be assessed using RECIST version 1.1.
Overall Survival (OS) | Up to 36 months
  OS is defined as the time from initiation of study treatment to death from any cause.
Number of participants experiencing any grade adverse events (AEs) as assessed by CTCAE v4.0 | Every 3 weeks during treatment, up to 24 months
  Adverse events will be collected and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Events of any grade will be recorded throughout the study.
Number of participants experiencing serious adverse events (SAEs) as defined by regulatory criteria | Throughout study participation, up to 24 months
  SAEs will be recorded and reported according to ICH and local regulatory definitions, including events such as death, life-threatening conditions, hospitalization, disability, or other medically significant events.
Change in quality of life measured by EORTC QLQ-C30 | Baseline and every 12 weeks, up to 24 months
  Quality of life will be assessed using the EORTC QLQ-C30, which evaluates global health status, five functional scales (physical, role, emotional, cognitive, and social), and multiple cancer-related symptoms (e.g., fatigue, pain, nausea).
  Scores range from 0 to 100. Higher scores on global health and functional scales indicate better functioning; higher scores on symptom scales indicate worse symptoms.
Change in hepatocellular carcinoma-specific quality of life measured by EORTC QLQ-HCC18 | Baseline and every 12 weeks, up to 24 months
  The EORTC QLQ-HCC18 will be used to assess liver cancer-specific symptoms and concerns, including fatigue, body image, nutrition, pain, jaundice, abdominal swelling, and fever.
  Each scale/item is scored from 0 to 100. Higher scores indicate worse symptoms or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Jyh Lin, Principal Investigator — National Cheng Kung University Hospital (NCKUH)
Locations (1):
- No. 138, Shengli Rd., North Dist, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matsui Y, Uhara J, Satoi S, Kaibori M, Yamada H, Kitade H, Imamura A, Takai S, Kawaguchi Y, Kwon AH, Kamiyama Y. Improved prognosis of postoperative hepatocellular carcinoma patients when treated with functional foods: a prospective cohort study. J Hepatol. 2002 Jul;37(1):78-86. doi: 10.1016/s0168-8278(02)00091-0. PMID 12076865
- [Result] Spierings EL, Fujii H, Sun B, Walshe T. A Phase I study of the safety of the nutritional supplement, active hexose correlated compound, AHCC, in healthy volunteers. J Nutr Sci Vitaminol (Tokyo). 2007 Dec;53(6):536-9. doi: 10.3177/jnsv.53.536. PMID 18202543
- [Result] Daddaoua A, Martinez-Plata E, Lopez-Posadas R, Vieites JM, Gonzalez M, Requena P, Zarzuelo A, Suarez MD, de Medina FS, Martinez-Augustin O. Active hexose correlated compound acts as a prebiotic and is antiinflammatory in rats with hapten-induced colitis. J Nutr. 2007 May;137(5):1222-8. doi: 10.1093/jn/137.5.1222. PMID 17449585
- [Result] Park HJ, Boo S, Park I, Shin MS, Takahashi T, Takanari J, Homma K, Kang I. AHCC(R), a Standardized Extract of Cultured Lentinula Edodes Mycelia, Promotes the Anti-Tumor Effect of Dual Immune Checkpoint Blockade Effect in Murine Colon Cancer. Front Immunol. 2022 Apr 20;13:875872. doi: 10.3389/fimmu.2022.875872. eCollection 2022. PMID 35514996

DOCUMENTS (1):
  • Study Protocol (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT07118735/Prot_000.pdf